CLINICAL TRIAL: NCT02221674
Title: Open-label Evaluation of the Population Pharmacokinetic Profile, Safety, Tolerability, and Efficacy of Tapentadol Oral Solution for the Treatment of Post-surgical Pain in Children Aged From Birth to Less Than 2 Years
Brief Title: Use of Tapentadol Oral Solution for Pain After Surgery in Children From Newborn to Less Than 2 Years Old
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Collaborators: Depomed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KF5503-72; 2014-000623-24 (EudraCT Number); U1111-1153-1662 (Other: WHO UTN); R331333PAI2007 (Other: Depomed Inc.)
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Moderate to Severe Acute Postoperative Pain
Keywords: Post-surgical pain; Opioid
MeSH Terms: conditions — Pain, Postoperative | interventions — Tapentadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tapentadol (Experimental): Tapentadol 4 mg/mL immediate release oral solution, single dose post-operatively.
  Interventions: Drug: Tapentadol

INTERVENTIONS:
Drug: Tapentadol
  Other Names: Palexia®; Nucynta®; Yantil®

SUMMARY:
This is a multicenter, open-label (all people involved know the identity of the intervention), single dose trial to evaluate the pharmacokinetic (PK) profile (how drugs are absorbed in the body, how are they distributed within the body and how are they removed from the body over time) in children aged from birth to less than 2 years after a surgical procedure that routinely produces moderate to severe acute post-surgical pain.

The trial will also evaluate the safety and tolerability of tapentadol oral solution in the population studied and the effect of tapentadol oral solution on pain.

DETAILED DESCRIPTION:
This clinical trial has 3 phases: enrollment, treatment (15 hours) and follow up.

During the enrolment phase consent and eligibility will be determined. After surgery, the participant will be given routine pain medication as per standard of care in the hospital.

Treatment phase: When the participant has a functioning gastrointestinal tract after surgery, can tolerate medication administered orally or via a feeding tube, meets the inclusion criteria, and does not meet any exclusion criterion, the participant will be allocated to the investigational medicinal product (IMP). Evaluations will be performed over the next 15 hours, including the assessment of the amount of pain. During this time, 2 blood samples will be taken for testing of the amount of tapentadol and its main metabolites in the participant's blood.

A final follow-up visit is planned to take place up to 2 weeks after taking the trial medication.

ELIGIBILITY:
Inclusion Criteria:

* The participant's parent(s) or legal guardian(s) have given written informed consent to participate.
* Participant is not obese (e.g., a body weight above the 97th percentile for children based on the World Health Organization weight charts) with a minimum body weight of 2.5 kg.
* Physical status rated not higher than P3 on the American Society of Anesthesiologists physical status classification in participants aged from 1 month to less than 2 years.
* Participant has undergone surgery that, in the investigator's opinion, would reliably produce moderate to severe pain requiring opioid treatment.
* At the time of allocation to IMP, participant has a sedation score that is not higher than 2 (moderately sedated) on the University of Michigan Sedation Scale with the exception of participants who are mechanically ventilated in age subgroup 3, has a functioning gastrointestinal tract after surgery, and can tolerate medication administered orally or via a feeding tube at the time of allocation to IMP.
* Participant has a reliable venous vascular access for pharmacokinetic blood sampling.

Exclusion Criteria:

* The participant's parent(s) or legal guardian(s) is an employee of the investigator or trial site, with direct involvement in this trial or other trials under the direction of that investigator or trial site, or the participant, or participant's parent(s), or legal guardian(s) is a family member of the employees or the investigator.
* Participant has been previously exposed to tapentadol.
* Participant has received an experimental drug or used an experimental medical device within 28 days before allocation to study medication, or within a period less than 10 times the drug's half-life, whichever is longer.
* Concomitant participation in another interventional clinical trial for the duration of this trial.
* Participant has undergone brain surgery.
* Participant has undergone a surgery that is expected to affect the absorption of tapentadol (e.g., to the gastrointestinal tract).
* Participant has a history or current condition of any one of the following:

  * Seizure disorder.
  * Traumatic or hypoxic brain injury, i.e. brain contusion, stroke, transient ischemic attack, intracranial bleeding or hematoma, brain neoplasm.
* Participant has a history or current condition of any one of the following:

  * Moderate to severe renal impairment.
  * Moderate to severe hepatic impairment, congestive hepatopathy, or hepatic portosystemic shunting.
  * Clinically relevant abnormal pulmonary function or clinically relevant respiratory disease that in the opinion of the investigator would put the participant at risk for developing respiratory depression, unless the participant is mechanically ventilated in age subgroup 3.
* Participant has signs or symptoms of congestive heart failure (e.g., requiring more than minimal inotropic support, an abnormal lactic acid value greater than 2-times upper limit of normal), or hemorrhagic disorder following surgery.
* Minimal inotropic medication is defined as:

  * Dopamine less or equal to 5 microgram/kg per minute.
  * Epinephrine less or equal to 0.03 microgram/kg per minute (but not both dopamine and epinephrine).
  * Milrinone less or equal to 0.5 microgram/kg per minute or less.
* Participant has a concomitant disease or disorder (e.g., endocrine, metabolic, neurological, or psychiatric disorder, or a febrile seizure or paralytic ileus) that in the opinion of the investigator may affect or compromise participant's safety during the trial participation.
* Participant has cognitive or developmental impairment such that trial participation may affect or compromise the participant's safety, or the participant's ability to comply with the protocol requirements (as appropriate for the participant's age), in the investigator's judgment. Otherwise, participant's with cognitive or developmental impairment may be enrolled in the trial.
* Participant has a clinically relevant history of hypersensitivity, allergy, or contraindication to tapentadol (or ingredients).
* Participant has:

  * Clinically relevant abnormal 12-lead ECG in the investigator's judgment.
  * Signs of pre-excitation syndrome.
  * Corrected QT (QTcF) interval greater than 460 ms. Participant may be allocated to Investigational Medicinal Product with values greater than 460 ms if, in the investigator's opinion, the value is a consequence of cardiac surgery and is not considered clinically significant.
* Participant has clinically relevant abnormal lab values from a sample obtained postoperatively and prior to allocation to study medication. The following specifications will apply:

  * Aspartate transaminase or alanine transaminase is greater than 2.5-times upper limit of normal.
  * Total bilirubin is greater than 2-times upper limit of normal and direct bilirubin is greater than 20% of the total bilirubin, and for participants in age subgroup 3, the presence of pathological jaundice in the opinion of the investigator.
  * Glomerular filtration rate (calculated according to Schwartz et al. 1984):
  * less than 20 mL/min/1.73 m2 for participants less than 1 week old.
  * less than 30 mL/min/1.73 m2 for participants 1 week to 8 weeks old.
  * less than 50 mL/min/1.73 m2 for participants more than 8 weeks old.
  * Other parameters (in the investigator's judgment).
* Signs or symptoms indicative of a systemic infection within 24 hours prior to allocation to study medication.
* Participant has been administered a prohibited medication.
* The mother of a newborn or the breastfeeding mother of a participant was administered a prohibited medication.
* At the time of dosing, in the investigator's judgment, the participant has either of the following:

  * Clinically unstable upper or lower airway conditions or respiratory depression (unless the participant is mechanically ventilated in age subgroup 3).
  * Clinically unstable systolic or diastolic blood pressure, heart rate, or respiratory rate.
* Participant has a peripheral oxygen saturation (SpO2) <92% for acyanotic participant, or <75% for cyanotic participant, with or without supplemental oxygen via nasal cannula or high flow nasal cannula, at the time of allocation to Investigational Medicinal Product.
* For age subgroup 1 and age subgroup 2, participant requires continuous positive airway pressure or mechanical ventilation, at the time of allocation to Investigational Medicinal Product.

Ages: 1 Day to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2016-10-14 (Actual); Study Completion 2016-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Director, Study Director — Grünenthal GmbH
Locations (7):
- United States (4):
  - US001, Palo Alto, California
  - US002, Louisville, Kentucky
  - US006, Durham, North Carolina
  - US004, Philadelphia, Pennsylvania
- Poland (2):
  - PL001, Lodz
  - PL004, Torun
- GB001, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Information available on the Grünenthal Group Web Site (see URL below for details); according to the European Federation of Pharmaceutical Industries and Associations (EFPIA) Data Sharing Principles.
URL: http://www.grunenthal.com/grt-web/Grunenthal_Group/Research_Development/Grunenthal_Clinical_Trials/Data_Sharing/296200025.jsp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient signed the informed consent on 05 Nov 2014. The last patient completed the trial on 03 Nov 2016. The trial followed a staggered recruitment by age, starting with the recruitment of patients in the oldest age group. Exposure and safety of at least 2 patients has been assessed before opening enrollment in the next younger age group.
Pre-assignment Details: Consent was obtained for 40 participants in the trial. 19 participants were allocated and received study drug (investigational medicinal product). Pharmacokinetic data was obtained for 18 participants.
  21 patients were enrolled but not allocated.
Groups:
- Participants Aged 6 Months to Less Than 2 Years: Infants aged 6 months to less than 2 years at the time of allocation to IMP (investigational medicinal product).
  Participants received a single dose of tapentadol oral solution postoperatively. The dose administered depended on the age of the subject and the body weight.
  Infants aged 6 months to less than 2 years received a dose of 0.75 mg/kg.
- Participants Aged 1 Month to Less Than 6 Months: Infants aged 1 month to less than 6 months at the time of allocation to IMP. Participants received a single dose of tapentadol oral solution postoperatively. The dose administered depended on the age of the subject and the body weight.
  Infants aged 1 month to less than 6 months received a dose of 0.60 mg/kg.
- Participants Aged From Birth to Less Than 1 Month: Neonates aged less than 1 month at the time of allocation to IMP (must be ≥37 weeks gestational age).
  Participants received a single dose of tapentadol oral solution postoperatively. The dose administered depended on the age of the subject and the body weight.
  Neonates aged less than 1 month received a dose of 0.50 mg/kg.
Period: Overall Study
Arm/Group | Participants Aged 6 Months to Less Than 2 Years | Participants Aged 1 Month to Less Than 6 Months | Participants Aged From Birth to Less Than 1 Month
Started | 8 | 6 | 5
Completed | 7 | 6 | 5
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is based on the participants allocated to IMP.
Groups:
- Participants Aged 6 Months to Less Than 2 Years: Infants aged 6 months to less than 2 years at the time of allocation to IMP. Participants received a single dose of tapentadol oral solution postoperatively. The dose administered depended on the age of the subject and the body weight.
  Infants aged 6 months to less than 2 years received a dose of 0.75 mg/kg.
- Total: Total of all reporting groups
Arm/Group | Participants Aged 6 Months to Less Than 2 Years | Participants Aged 1 Month to Less Than 6 Months | Participants Aged From Birth to Less Than 1 Month | Total
Number analyzed (Participants) | 8 | 6 | 5 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 6 | 5 | 19
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 420.0 (147.8) | 92.8 (37.9) | 14.6 (8.5) | 210.0 (209.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 3 | 9
  Male | 4 | 4 | 2 | 10
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 2 | 15
  Poland | 0 | 0 | 3 | 3
  United Kingdom | 1 | 0 | 0 | 1
Height [Mean (Standard Deviation); unit: centimeter] | 73.3 (5.2) | 62.0 (4.3) | 53.4 (4.4) | 64.5 (9.5)
Weight [Mean (Standard Deviation); unit: kilogram] | 9.21 (1.50) | 5.92 (1.18) | 3.78 (0.66) | 6.74 (2.59)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter] | 17.11 (1.36) | 15.28 (1.31) | 13.36 (2.49) | 15.55 (2.24)
Baseline Pain Intensity using the FLACC Scale [Mean (Standard Deviation); unit: units on a scale] — Pain intensity using the Face, Legs, Activity, Cry, Consolability Scale (FLACC Scale) at baseline visit.
  The FLACC Scale is a behavioral scale for scoring postoperative pain in young children. It includes five categories of pain behaviors, including facial expression, leg movement, activity, cry, and consolability. The scale is scored in a range of 0-10 with 0 representing no pain.
  units on a scale | 2.8 (2.9) | 3.8 (3.9) | 1.6 (1.5) | 2.8 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Evaluation Based on Serum Concentrations of Tapentadol After a Single Dose of Tapentadol Oral Solution in Participants Aged 6 Months to Less Than 2 Years
Description: The pharmacokinetic profile of Tapentadol and its major metabolite tapentadol-O-glucuronide was evaluated to enable data based recommendations for the use of Tapentadol in children of different ages.
  Each participant had a single pharmacokinetic sample taken at up to 2 different pre-defined time points.
  Serum was analyzed using liquid chromatography-tandem mass spectrometry. Mean and Standard Deviation of Serum Concentrations of Tapentadol were calculated.
  Summary statistics at a given time point were only determined if at least 2 participants had observations above the lower limit of quantification (LLOQ).
  If overall only a single sample was available at one of the pre-defined time points, the measured value is presented and the standard deviation is given as N/A.
Time Frame: Up to 8 hours after IMP administration
Population: The trial used sparse sampling for the assessment of Pharmacokinetic. Overall, there were 6 time points for sampling. Participants were allocated to 2 different time points for a blood sample to be taken. Some participants only had one sample taken. Some samples were below the Lower limit of quantification (LLOQ).
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Groups:
- Participants Aged 6 Months to Less Than 2 Years - PK Set: Infants aged 6 months to less than 2 years at the time of allocation to IMP who had quantifiable serum concentrations.
Arm/Group | Participants Aged 6 Months to Less Than 2 Years - PK Set
Number analyzed (Participants) | 7
nanogram per milliliter
  30 minutes after administration: number analyzed (Participants) | 3
  30 minutes after administration | 9.8 (5.21)
  1 hour after administration: number analyzed (Participants) | 1
  1 hour after administration | 18.79 (NA) — One sample was used at this specified time point.
  2 hours after administration: number analyzed (Participants) | 2
  2 hours after administration | 32.2 (14.92)
  4 hours after administration: number analyzed (Participants) | 3
  4 hours after administration | 11.1 (5.97)
  6 hours after administration: number analyzed (Participants) | 1
  6 hours after administration | 14.85 (NA) — One sample was used at this specified time point.
  8 hours after administration: number analyzed (Participants) | 2
  8 hours after administration | 10.7 (4.15)

2. Primary Outcome: Pharmacokinetic Evaluation Based on Serum Concentrations of Tapentadol After a Single Dose of Tapentadol Oral Solution in Participants Aged 1 Month to Less Than 6 Months
Description: as for outcome 1
Time Frame: Up to 8 hours after IMP administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Groups:
- Participants Aged 1 Month to Less Than 6 Months - PK Set: Infants aged 1 month to less than 6 months at the time of allocation to IMP who had quantifiable serum concentrations.
Arm/Group | Participants Aged 1 Month to Less Than 6 Months - PK Set
Number analyzed (Participants) | 6
nanogram per milliliter
  30 minutes after administration: number analyzed (Participants) | 2
  30 minutes after administration | 8.3 (6.30)
  1 hour after administration: number analyzed (Participants) | 1
  1 hour after administration | 35.27 (NA) — One sample was used at this specified time point.
  2 hours after administration: number analyzed (Participants) | 3
  2 hours after administration | 27.3 (0.81)
  4 hours after administration: number analyzed (Participants) | 2
  4 hours after administration | 25.9 (10.33)
  6 hours after administration: number analyzed (Participants) | 1
  6 hours after administration | 32.75 (NA) — One sample was used at this specified time point.
  8 hours after administration: number analyzed (Participants) | 2
  8 hours after administration | 5.6 (1.81)

3. Primary Outcome: Pharmacokinetic Evaluation Based on Serum Concentrations of Tapentadol After a Single Dose of Tapentadol Oral Solution in Participants Aged From Birth to Less Than 1 Month
Description: as for outcome 1
Time Frame: Up to 8 hours after IMP
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Groups:
- Participants Aged From Birth to Less Than 1 Month - PK Set: Neonates aged less than 1 month (must be ≥37 weeks gestational age) at the time of allocation to IMP who had quantifiable serum concentrations.
Arm/Group | Participants Aged From Birth to Less Than 1 Month - PK Set
Number analyzed (Participants) | 5
nanogram per milliliter
  30 minutes after administration: number analyzed (Participants) | 1
  30 minutes after administration | 26.62 (NA) — One sample was used at this specified time point.
  1 hour after administration: number analyzed (Participants) | 1
  1 hour after administration | 43.63 (NA) — One sample was used at this specified time point.
  2 hours after administration: number analyzed (Participants) | 2
  2 hours after administration | 19.9 (7.67)
  4 hours after administration: number analyzed (Participants) | 2
  4 hours after administration | 15.0 (8.92)
  6 hours after administration: number analyzed (Participants) | 1
  6 hours after administration | 18.82 (NA) — One sample was used at this specified time point.
  8 hours after administration: number analyzed (Participants) | 2
  8 hours after administration | 14.6 (6.26)

4. Primary Outcome: Pharmacokinetic Profile of Serum Concentrations of Tapentadol-O-glucuronide After a Single Dose of Tapentadol Oral Solution in Participants Aged 6 Months to Less Than 2 Years
Description: The pharmacokinetic profile of Tapentadol and its major metabolite tapentadol-O-glucuronide was evaluated to enable data based recommendations for the use of Tapentadol in children of different ages.
  Each participant had a single pharmacokinetic sample taken at up to 2 different pre-defined time points.
  Serum was analyzed using liquid chromatography-tandem mass spectrometry. Mean and Standard Deviation of Serum Concentrations of tapentadol-O-glucuronide were calculated.
  Summary statistics at a given time point were only determined if at least 2 participants had observations above the lower limit of quantification (LLOQ).
  If overall only a single sample was available at one of the pre-defined time points, the measured value is presented and the standard deviation is given as N/A.
Time Frame: Up to 8 hours after IMP
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Participants Aged 6 Months to Less Than 2 Years - PK Set
Number analyzed (Participants) | 7
nanogram per milliliter
  30 minutes after administration: number analyzed (Participants) | 3
  30 minutes after administration | 105.7 (125.00)
  1 hour after administration: number analyzed (Participants) | 1
  1 hour after administration | 430.7 (NA) — One sample was used at this specified time point.
  2 hours after administration: number analyzed (Participants) | 2
  2 hours after administration | 468.0 (248.41)
  4 hours after administration: number analyzed (Participants) | 3
  4 hours after administration | 348.7 (228.22)
  6 hours after administration: number analyzed (Participants) | 1
  6 hours after administration | 370.2 (NA) — One sample was used at this specified time point.
  8 hours after administration: number analyzed (Participants) | 2
  8 hours after administration | 285.1 (107.06)

5. Primary Outcome: Pharmacokinetic Profile of Serum Concentrations of Tapentadol-O-glucuronide After a Single Dose of Tapentadol Oral Solution in Participants Aged 1 Month to Less Than 6 Months
Description: as for outcome 4
Time Frame: Up to 8 hours after IMP
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Participants Aged 1 Month to Less Than 6 Months - PK Set
Number analyzed (Participants) | 6
nanogram per milliliter
  30 minutes after administration: number analyzed (Participants) | 1
  30 minutes after administration | 128.8 (NA) — One sample was used at this specified time point.
  1 hour after administration: number analyzed (Participants) | 1
  1 hour after administration | 136.3 (NA) — One sample was used at this specified time point.
  2 hours after administration: number analyzed (Participants) | 3
  2 hours after administration | 324.9 (116.61)
  4 hours after administration: number analyzed (Participants) | 2
  4 hours after administration | 449.7 (7.42)
  6 hours after administration: number analyzed (Participants) | 1
  6 hours after administration | 253.3 (NA) — One sample was used at this specified time point.
  8 hours after administration: number analyzed (Participants) | 2
  8 hours after administration | 92.2 (63.83)

6. Primary Outcome: Pharmacokinetic Profile of Serum Concentrations of Tapentadol-O-glucuronide After a Single Dose of Tapentadol Oral Solution in Participants Aged From Birth to Less Than 1 Month
Description: as for outcome 4
Time Frame: Up to 8 hours after IMP
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Participants Aged From Birth to Less Than 1 Month - PK Set
Number analyzed (Participants) | 5
nanogram per milliliter
  30 minutes after administration: number analyzed (Participants) | 1
  30 minutes after administration | 74.38 (NA) — One sample was used at this specified time point.
  1 hour after administration: number analyzed (Participants) | 1
  1 hour after administration | 209 (NA) — One sample was used at this specified time point.
  2 hours after administration: number analyzed (Participants) | 2
  2 hours after administration | 98.5 (2.62)
  4 hours after administration: number analyzed (Participants) | 2
  4 hours after administration | 147.6 (53.74)
  6 hours after administration: number analyzed (Participants) | 1
  6 hours after administration | 224.8 (NA) — One sample was used at this specified time point.
  8 hours after administration: number analyzed (Participants) | 2
  8 hours after administration | 174.1 (11.03)

7. Other Pre Specified Outcome: Change From Baseline (Visit 1, After Surgery) in Pain Intensity
Description: The change from baseline in pain intensity using the Face, Legs, Activity, Cry, Consolability Scale (FLACC Scale) at 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, and 15 hours after a single dose of tapentadol.
  The FLACC Scale is a behavioral scale for scoring postoperative pain in young children. It includes five categories of pain behaviors, including facial expression, leg movement, activity, cry, and consolability. The scale is scored in a range of 0-10 with 0 representing no pain.
  The pain intensity scores were summarized descriptively per scheduled time point.
Time Frame: Baseline; up to 15 hours after study medication
Population: For the Arm/Group "Participants aged 6 months to less than 2 years" only 7 values were available at the timepoint "6 hours after administration".
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Aged 6 Months to Less Than 2 Years. | Participants Aged 1 Month to Less Than 6 Months. | Participants Aged From Birth to Less Than 1 Month.
Number analyzed (Participants) | 8 | 6 | 5
units on a scale
  15 minutes after administration | -0.8 (3.1) | -1.3 (2.8) | -1.6 (1.5)
  30 minutes after administration | -1.1 (2.6) | -3.0 (3.6) | -1.4 (1.5)
  1 hour after administration | -2.0 (3.6) | -2.7 (4.5) | 0.0 (3.7)
  2 hours after administration | -2.8 (2.9) | -3.0 (3.9) | -0.4 (2.6)
  4 hours after administration | -1.6 (3.4) | -2.2 (3.3) | -0.4 (2.3)
  6 hours after administration: number analyzed (Participants) | 7 | 6 | 5
  6 hours after administration | -1.9 (3.1) | -1.7 (4.8) | -0.4 (2.3)
  8 hours after administration | -2.5 (2.5) | -3.0 (3.2) | -1.2 (1.1)
  12 hours after administration | -2.4 (2.8) | -3.5 (3.8) | -1.4 (1.5)
  15 hours after administration | -2.1 (3.5) | -3.8 (3.9) | -1.0 (2.1)

ADVERSE EVENTS:
Time Frame: Any Adverse Events (AE) that started on the intake of the IMP (investigational medicinal product) up to the end of the therapeutic reach of the IMP. Any pre-treatment AE which worsened (change in intensity, frequency or quality) after IMP administration compared to the complaint present before IMP intake have been recorded as a new AE.
Description: The therapeutic reach is the time after IMP intake that a subject is still considered to be potentially affected by a study drug. For tapentadol oral solution, the therapeutic reach is defined as 48 hours after (last) IMP intake.
Arm/Group | Participants Aged 6 Months to Less Than 2 Years. | Participants Aged 1 Month to Less Than 6 Months. | Participants Aged From Birth to Less Than 1 Month.
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 3/8 | 3/6 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Aged 6 Months to Less Than 2 Years. (N=8) | Participants Aged 1 Month to Less Than 6 Months. (N=6) | Participants Aged From Birth to Less Than 1 Month. (N=5)
Junctional ectopic tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (2)
Stoma site erythema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 1 (3)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right to review any publication pertaining to the trial before it is submitted for publication. Neither party has the right to prohibit publication unless publication can be shown to affect possible patent rights.